CLINICAL TRIAL: NCT05857462
Title: A Randomized Controlled Trial to Evaluate the Impact of Integrated Preoperative Fascia Iliaca Compartment Block (FICB) for Fast-track Surgery in Elderly Hip Fracture
Brief Title: The Impact of Integrated Preoperative Fascia Iliaca Compartment Block in Elderly Hip Fracture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Ministry of Health, Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CREC015/2023
Record Dates: First submitted 2023-03-29; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Hip Fractures; Pain, Acute; Hip Fracture Surgery; Delirium in Old Age; Pain Intensity
MeSH Terms: conditions — Hip Fractures; Acute Pain; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post-admission FICB (Experimental): Post-admission FICB, drug 0.33% bupivacaine 30 ml + Pre-operative FICB 0.33% bupivacaine 30 ml. Peri-operative pain management protocol : paracetamol + opioid.
  Interventions: Procedure: Post-admission FICB
- Only preoperative FICB (No Intervention): No post-admission FICB + Pre-operative FICB 0.33% bupivacaine 30 ml. Peri-operative pain management protocol : paracetamol + opioid.

INTERVENTIONS:
Procedure: Post-admission FICB — Post-admission supra-inguinal FICB in hip fracture patient with 0.33% bupivacaine 30 ml
  Arms: Post-admission FICB

SUMMARY:
This prospective randomized controlled study is aimed to determine the advantages of post-admission fascia iliaca compartment block (FICB) in geriatric hip fracture surgery combination with multimodal analgesia compared with no post-admission FICB. The primary outcome is incidence of delirium during hospital admission. Secondary outcomes are incidence of delirium at hospital discharge, pre- and post-operative pain intensity, peri-operative complications, opioid-related side effects, post-operative complications and length of hospital stay, and morbidities and mortality (in-hospital and 30 days).

DETAILED DESCRIPTION:
Population: elderly patients age ≥ 65 years old, diagnosed with an isolated acute hip fracture within 7 days and plan to receive fast-track hip fracture. Statistic analysis plan surgery within 48 hours after hospital admission.

Study population: elderly isolated hip fracture patients who are admitted in those 8 hospitals centers in Thailand and have moderate pain or higher than moderate pain during movement since hospital admission.

Sample size : 210 patients per group (drop out 10%) total 420 patients

Statistical analysis: SPSS will be used for study analysis. The category variables will be present as number and percentage, and chi-square or fisher exact test will be used to compare between the groups.The continuous variables will be tested the distribution, data presentation will be mean and standard deviation (SD) for normal distribution while median and interquartile rang (IQR) for non-normal distribution. Student t test or Wilcoxson rank some test will be used as appropriate to test for different between the group. And p value less than 0.05 will be considered statically significance.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are aged ≥65 , <85 years old and diagnose hip fracture in 8 hospitals
2. Planed for fast-track hip surgery
3. Isolated acute hip fracture
4. Pain on admission during movement ≥ 4 (moderate pain)

Exclusion Criteria:

1. refusal to participate the study
2. ASA physical status >III

2. duration of fracture more than 7 days before admission 3. hip fracture after/at previous instrumentation 4. hip fracture causing by a traffic accident or high energy force 5. suspected pathologic fracture 6. unable to communication 7. abnormal consciousness or severe cognitive dysfunction that could not communication such as mental retardation, severe Alzheimer's disease and schizophenia 8. allergy to local anesthetic drug

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
In-hospital Delirium | In hospital admission, assess up to 30 days
  Incidence of delirium using Nursing Delirium Screening Scale (NU-DESC) Thai version plus backward counting 30-1. Total Scale 11 ( > or = 2 means delirium). The patient will be assessed once a day in the morning period.

SECONDARY OUTCOMES:
Preoperative pain score | 48 hours after hospital admission
  Numeric rating scale (0-10; 0=no pain, 10 worst pain imaginable) will be used. The patient will be assessed every 6 hours duration until receiving surgery within 48 hours.
Post-operative pain score | Until postoperative 72 hours
  Numeric rating scale (0-10; 0=no pain, 10 worst pain imaginable) will be used. The patient will be assessed every 6 hours duration postoperatively until 72 hours
Preoperative morphine consumption | 48 hours after hospital admission
  Milligram morphine equivalent
Postoperative morphine consumption | Until postoperative 72 hours
  Milligram morphine equivalent
Major adverse cardiac events | In hospital admission, up to 30 days
  Incidence of major adverse cardiac events (fatal arrythmia, cardiac arrest, myocardial infarction, stroke, pulmonary emboli)
In-hospital morbidities | In hospital admission, up to 30 days
  Incidence of in-hospital morbidities include deep vein thrombosis sepsis, pneumonia, respiratory failure, urinary tract infection, acute kidney injury
Discharge hospital status | On hospital discharge day, up to 30 days
  Self-care ability to perform the activity of daily living (ADLs)
Length of hospital stay | In hospital admission, up to 30 days
  Days of hospital stay
In-hospital mortality rate | In hospital admission, up to 30 days
  Incidence related to all causes of death implant related (implant removal, implant exchange, implant failure,) infection related, bleeding related, non-union fracture, re-fracture
30 days mortality | In hospital admission, up to 30 days
  Incidence of death
Predict 30-day mortality in hip fracture patient with multiple comorbidities | On admission day
  Charlson Comorbidity Index (CCI) with 19 item-version (adjusted weights for each condition). Higher score of Charlson Comorbidity Index (CCI) is related to higher mortality. CCI score 1-2 = mild, 3-5 scores = moderate, > or = 5 scores = severe.

CONTACTS AND LOCATIONS:
Overall Officials: Suwimon Tangwiwat, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chotanaphuti T, Jareonarpornwatana A, Laoruengthana A. The mortality rate after thromboembolism prophylaxis in the hip fracture surgery. J Med Assoc Thai. 2009 Dec;92 Suppl 6:S115-9. PMID 20120672
- [Background] Chaysri R, Leerapun T, Klunklin K, Chiewchantanakit S, Luevitoonvechkij S, Rojanasthien S. Factors related to mortality after osteoporotic hip fracture treatment at Chiang Mai University Hospital, Thailand, during 2006 and 2007. J Med Assoc Thai. 2015 Jan;98(1):59-64. PMID 25775733
- [Background] Kulachote N, Sa-Ngasoongsong P, Sirisreetreerux N, Wongsak S, Suphachatwong C, Wajanavisit W, Kawinwonggowit V. The Impacts of Early Hip Surgery in High-Risk Elderly Taking Antithrombotic Agents and Afflicted with Intertrochanteric Fracture. J Med Assoc Thai. 2015 Sep;98 Suppl 8:S76-81. PMID 26529819
- [Background] Haugan K, Johnsen LG, Basso T, Foss OA. Mortality and readmission following hip fracture surgery: a retrospective study comparing conventional and fast-track care. BMJ Open. 2017 Aug 29;7(8):e015574. doi: 10.1136/bmjopen-2016-015574. PMID 28851773
- [Background] Pollmann CT, Rotterud JH, Gjertsen JE, Dahl FA, Lenvik O, Aroen A. Fast track hip fracture care and mortality - an observational study of 2230 patients. BMC Musculoskelet Disord. 2019 May 24;20(1):248. doi: 10.1186/s12891-019-2637-6. PMID 31122228
- [Background] Munoz Vives JM, Jornet-Gibert M, Camara-Cabrera J, Esteban PL, Brunet L, Delgado-Flores L, Camacho-Carrasco P, Torner P, Marcano-Fernandez F; Spanish HIP-COVID Investigation Group. Mortality Rates of Patients with Proximal Femoral Fracture in a Worldwide Pandemic: Preliminary Results of the Spanish HIP-COVID Observational Study. J Bone Joint Surg Am. 2020 Jul 1;102(13):e69. doi: 10.2106/JBJS.20.00686. PMID 32618917
- [Background] Lewis PM, Waddell JP. When is the ideal time to operate on a patient with a fracture of the hip? : a review of the available literature. Bone Joint J. 2016 Dec;98-B(12):1573-1581. doi: 10.1302/0301-620X.98B12.BJJ-2016-0362.R2. PMID 27909117
- [Background] Pincus D, Ravi B, Wasserstein D, Huang A, Paterson JM, Nathens AB, Kreder HJ, Jenkinson RJ, Wodchis WP. Association Between Wait Time and 30-Day Mortality in Adults Undergoing Hip Fracture Surgery. JAMA. 2017 Nov 28;318(20):1994-2003. doi: 10.1001/jama.2017.17606. PMID 29183076
- [Background] Jiang M, Liu S, Deng H, Liang X, Bo Z. The efficacy and safety of fast track surgery (FTS) in patients after hip fracture surgery: a meta-analysis. J Orthop Surg Res. 2021 Feb 27;16(1):162. doi: 10.1186/s13018-021-02277-w. PMID 33639957
- [Background] Steenberg J, Moller AM. Systematic review of the effects of fascia iliaca compartment block on hip fracture patients before operation. Br J Anaesth. 2018 Jun;120(6):1368-1380. doi: 10.1016/j.bja.2017.12.042. Epub 2018 Apr 5. PMID 29793602
- [Background] Fadhlillah F, Chan D, Pelosi P, Rubulotta F. Systematic review and meta-analysis of single injection fascia iliaca blocks in the peri-operative management of patients with hip fractures. Minerva Anestesiol. 2019 Nov;85(11):1211-1218. doi: 10.23736/S0375-9393.19.13535-3. Epub 2019 Jul 4. PMID 31274264
- [Background] Wan HY, Li SY, Ji W, Yu B, Jiang N. Fascia Iliaca Compartment Block for Perioperative Pain Management of Geriatric Patients with Hip Fractures: A Systematic Review of Randomized Controlled Trials. Pain Res Manag. 2020 Nov 25;2020:8503963. doi: 10.1155/2020/8503963. eCollection 2020. PMID 33294087
- [Background] Hao J, Dong B, Zhang J, Luo Z. Pre-emptive analgesia with continuous fascia iliaca compartment block reduces postoperative delirium in elderly patients with hip fracture. A randomized controlled trial. Saudi Med J. 2019 Sep;40(9):901-906. doi: 10.15537/smj.2019.9.24483. PMID 31522217
- [Background] Foss NB, Kristensen BB, Bundgaard M, Bak M, Heiring C, Virkelyst C, Hougaard S, Kehlet H. Fascia iliaca compartment blockade for acute pain control in hip fracture patients: a randomized, placebo-controlled trial. Anesthesiology. 2007 Apr;106(4):773-8. doi: 10.1097/01.anes.0000264764.56544.d2. PMID 17413915
- [Background] Groot L, Dijksman LM, Simons MP, Zwartsenburg MM, Rebel JR. Single Fascia Iliaca Compartment Block is Safe and Effective for Emergency Pain Relief in Hip-fracture Patients. West J Emerg Med. 2015 Dec;16(7):1188-93. doi: 10.5811/westjem.2015.10.28270. Epub 2015 Dec 14. PMID 26759680
- [Background] Diakomi M, Papaioannou M, Mela A, Kouskouni E, Makris A. Preoperative fascia iliaca compartment block for positioning patients with hip fractures for central nervous blockade: a randomized trial. Reg Anesth Pain Med. 2014 Sep-Oct;39(5):394-8. doi: 10.1097/AAP.0000000000000133. PMID 25068412
- [Background] Kacha NJ, Jadeja CA, Patel PJ, Chaudhari HB, Jivani JR, Pithadia VS. Comparative Study for Evaluating Efficacy of Fascia Iliaca Compartment Block for Alleviating Pain of Positioning for Spinal Anesthesia in Patients with Hip and Proximal Femur Fractures. Indian J Orthop. 2018 Mar-Apr;52(2):147-153. doi: 10.4103/ortho.IJOrtho_298_16. PMID 29576642
- [Background] Hsu YP, Hsu CW, Bai CH, Cheng SW, Chen C. Fascia iliaca compartment block versus intravenous analgesic for positioning of femur fracture patients before a spinal block: A PRISMA-compliant meta-analysis. Medicine (Baltimore). 2018 Dec;97(49):e13502. doi: 10.1097/MD.0000000000013502. PMID 30544447
- [Background] Nie H, Yang YX, Wang Y, Liu Y, Zhao B, Luan B. Effects of continuous fascia iliaca compartment blocks for postoperative analgesia in patients with hip fracture. Pain Res Manag. 2015 Jul-Aug;20(4):210-2. doi: 10.1155/2015/872651. Epub 2015 Jun 30. PMID 26125194
- [Background] Lawlor PG, Bush SH. Delirium diagnosis, screening and management. Curr Opin Support Palliat Care. 2014 Sep;8(3):286-95. doi: 10.1097/SPC.0000000000000062. PMID 25004177
- [Background] Li H, Zheng ZN, Zhang NR, Guo J, Wang K, Wang W, Li LG, Jin J, Tang J, Liao YJ, Jin SQ. Intra-operative open-lung ventilatory strategy reduces postoperative complications after laparoscopic colorectal cancer resection: A randomised controlled trial. Eur J Anaesthesiol. 2021 Oct 1;38(10):1042-1051. doi: 10.1097/EJA.0000000000001580. PMID 34366425
- [Background] Fixation using Alternative Implants for the Treatment of Hip fractures (FAITH) Investigators. Fracture fixation in the operative management of hip fractures (FAITH): an international, multicentre, randomised controlled trial. Lancet. 2017 Apr 15;389(10078):1519-1527. doi: 10.1016/S0140-6736(17)30066-1. Epub 2017 Mar 3. PMID 28262269
- [Background] Mouzopoulos G, Vasiliadis G, Lasanianos N, Nikolaras G, Morakis E, Kaminaris M. Fascia iliaca block prophylaxis for hip fracture patients at risk for delirium: a randomized placebo-controlled study. J Orthop Traumatol. 2009 Sep;10(3):127-33. doi: 10.1007/s10195-009-0062-6. Epub 2009 Aug 19. PMID 19690943
- See also: National Institute for Health and Care Excellence. Clinical guideline: Hip fracture: management 2011. — http://www.nice.org.uk/guidance/cg124